CLINICAL TRIAL: NCT01333007
Title: A Cohort Study of First-line Treatment of Patients With Unresectable Advanced (Stage IIIB), Metastatic (Stage IV) or Recurrent Non Squamous Non-small Cell Lung Cancer (NSCLC), Starting a Treatment With Bevacizumab (Avastin®) in Combination With Chemotherapy.
Brief Title: An Observational Study of Avastin (Bevacizumab) in Combination With Chemotherapy in Patients With Metastatic or Recurrent Non-Squamous Non-Small Cell Lung Cancer
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML22991
Record Dates: First submitted 2011-04-06; First posted 2011-04-11 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Non-Squamous Non-Small Cell Lung Cancer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Cohort

SUMMARY:
This observational study will evaluate modality, efficacy and safety of Avastin (bevacizumab) as first-line treatment in combination with chemotherapy in patients with inoperable advanced, metastatic or recurrent non-squamous non-small cell lung cancer in clinical practice. Data will be collected for each patient for 18 months from initiation of Avastin therapy.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, >/= 18 years of age
* Inoperable advanced, metastatic or recurrent non-squamous non-small cell lung cancer (NSCLC)
* Treating physician's decision to initiate first-line Avastin treatment

Exclusion Criteria:

* Participation in a clinical trial evaluating anti-cancer therapies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients With Metastatic or Recurrent Non-Squamous Non-Small Cell Lung Cancer
Sampling Method: Probability Sample
Enrollment: 423 (Actual)
Dates: Start 2010-07; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Progression-free survival | 18 months

SECONDARY OUTCOMES:
Clinical (diagnosis, therapies, comorbidity) and demographic characteristics of patients initiated on Avastin treatment | 18 months
Modality of treatment with Avastin (dose, duration, associated chemotherapy) | 18 months
Overall survival | 18 months
Safety: Incidence of adverse events | 18 months
Quality of Life: Functional Assessment of Cancer Therapy-Lung (FACT-L) questionnaire | 18 months
Treatment of non-squamous NSCLC in clinical practice | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (127):
- France (127):
  - Abbeville
  - Agen
  - Aix-en-Provence
  - Alès
  - Ambilly
  - Amiens
  - Amilly
  - Angers
  - Annecy
  - Antibes
  - Armentières
  - Arras
  - Aubenas
  - Aulnay-sous-Bois
  - Auxerre
  - Bar-le-Duc
  - Bastia
  - Bayeux
  - Bayonne
  - Besançon
  - Beuvry
  - Biarritz
  - Bobigny
  - Bois-Guillaume
  - Bordeaux
  - Boulogne-sur-Mer
  - Bourg-en-Bresse
  - Brest
  - Brive-la-Gaillarde
  - Bron
  - Bry-sur-Marne
  - Caen
  - Cagnes-sur-Mer
  - Cahors
  - Carcassonne
  - Chalon-sur-Saône
  - Chambray-lès-Tours
  - Charleville-Mézières
  - Chaumont
  - Chauny
  - Châteauroux
  - Cherbourg Octeville
  - Clamart
  - Clermont-Ferrand
  - Colmar
  - Compiègne
  - Cornebarrieu
  - Creil
  - Créteil
  - Dax
  - Dijon
  - Dunkirk
  - Eaubonne
  - Épernay
  - Évreux
  - Fontainebleau
  - Gap
  - Gleizé
  - Granville
  - Hyères
  - La Chaussée-Saint-Victor
  - La Roche-sur-Yon
  - La Seyne-sur-Mer
  - La Source
  - Le Mans
  - Le Perreux-sur-Marne
  - Levallois-Perret
  - Libourne
  - Liévin
  - Lille
  - Limoges
  - Longjumeau
  - Lorient
  - Lormont
  - Lyon
  - Mareuil-lès-Meaux
  - Marseille
  - Maubeuge
  - Meaux
  - Metz
  - Metz-Tessy
  - Mont-de-Marsan
  - Montauban
  - Montélimar
  - Montfermeil
  - Montpellier
  - Mulhouse
  - Nancy
  - Narbonne
  - Nemours
  - Neuilly-sur-Seine
  - Nevers
  - Osny
  - Paris
  - Pau
  - Perpignan
  - Pierre-Bénite
  - Pontarlier
  - Pontoise
  - Rambouillet
  - Reims
  - Rennes
  - Rouen
  - Saint-Aubin-lès-Elbeuf
  - Saint-Herblain
  - Saint-Jean
  - Saint-Lô
  - Saint-Priest-en-Jarez
  - Saint-Quentin
  - Saintes
  - Senlis
  - Soissons
  - Ste Feyre
  - Strasbourg
  - Tarbes
  - Thionville
  - Thonon-les-Bains
  - Toulon
  - Toulouse
  - Vandœuvre-lès-Nancy
  - Vannes
  - Verdun
  - Versailles
  - Vesoul
  - Vénissieux
  - Vichy
  - Villeneuve-Saint-Georges